CLINICAL TRIAL: NCT05344287
Title: The Impact of a Plant-Based Diet on Indices of Cardiovascular Health in African Americans: A Cross-Sectional Study
Brief Title: Impact of a Plant-Based Diet on Indices of Cardiovascular Health in African Americans
Status: Completed | Type: Observational
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Associate Professor, The University of Texas at Arlington
Other Study IDs: 2019-0318
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Diseases; Hypertension; Diet, Healthy
Keywords: health disparity; endothelial function; hypertension; vegan diet; Black Americans; inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Inflammation | interventions — Diet, Plant-Based

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — stored serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typical American Diet: African American individuals who self-report adhering to a typical American diet prior to enrolling in the study.
  Interventions: Other: Typical American Diet
- Plant-Based Diet: African American individuals who self-report adhering to a plant-based diet prior to enrolling in the study.
  Interventions: Other: Plant-Based Diet

INTERVENTIONS:
Other: Typical American Diet — Participants self-reported adherence to a typical American diet prior to enrolling in the study. This factor determined cross-sectional group allocation.
  Groups: Typical American Diet
Other: Plant-Based Diet — Participants self-reported adherence to a 100% plant-based diet prior to enrolling in the study. This factor determined cross-sectional group allocation.
  Groups: Plant-Based Diet

SUMMARY:
The role of diet in preventing hypertension and cardiovascular diseases in African Americans, who have a much higher risk of developing these diseases, is not well understood. Therefore, this project will investigate whether African Americans following a 100% plant-based diet have more optimal blood pressure, vascular function, and blood lipid profiles, along with lower systemic inflammation relative to African Americans following a typical American diet.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American/Black
* Self-reported adherence to either a typical American diet (not following a specific diet pattern) or 100% plant-based (vegan) diet
* Age 18-40

Exclusion Criteria:

* History of smoking within 2 years or being a current smoker
* Taking vasoactive medications
* Having overt cardiovascular, metabolic, or neurological disease
* Pregnant individuals

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample from the greater Dallas-Fort Worth Metroplex area.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Lipid profile (Total-C, LDL-C, VLDL-C, HDL-C, TG) | Day 1
C-reactive protein | Day 1
Post-occlusive brachial artery flow-mediated dilation (% change in brachial artery diameter from resting baseline) | Day 1
Post-occlusive forearm reactive hyperemia (% change in brachial artery blood velocity from resting baseline) | Day 1
Pulse wave velocity (carotid-to-femoral) | Day 1
Augmentation index (AIx@HR75) | Day 1
Cerebral vascular reactivity (% change in cerebrovascular conductance index from resting baseline) | Day 2
Local cutaneous thermal hyperemia (% change in cutaneous vascular conductance from resting baseline) | Day 2
Peripheral blood pressure (systolic, diastolic, mean) | Day 1
Central blood pressure (systolic, diastolic, mean) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Brothers, PhD, Principal Investigator — The University of Texas at Arlington
Locations (1):
- UT Arlington - Science and Engineering Innovation and Research Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data Availability Statement: All raw data were collected and generated at the University of Texas at Arlington. Data supporting the findings and conclusions of this study are available from the corresponding author upon request.

REFERENCES:
- [Derived] Martin ZT, Olvera G, Villegas CA, Campbell JC, Akins JD, Brown KK, Brothers RM. The impact of a plant-based diet on indices of cardiovascular health in African Americans: a cross-sectional study. Appl Physiol Nutr Metab. 2022 Sep 1;47(9):903-914. doi: 10.1139/apnm-2022-0027. Epub 2022 May 5. PMID 35512369